CLINICAL TRIAL: NCT00461292
Title: Safety and Efficacy Study of Botulinum Toxin Type A for the Treatment of Neurogenic Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-516
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): botulinum toxin Type A (200U)
  Interventions: Biological: botulinum toxin Type A (200U)
- 2 (Experimental): botulinum toxin Type A (300U)
  Interventions: Biological: botulinum toxin Type A (300U)
- 3 (Other): placebo; botulinum toxin Type A (200U)
  Interventions: Other: Normal saline (Placebo); botulinum toxin Type A (200U)
- 4 (Other): placebo; botulinum toxin Type A (300U)
  Interventions: Other: Normal saline (Placebo); botulinum toxin Type A (300U)

INTERVENTIONS:
Biological: botulinum toxin Type A (200U) — botulinum toxin Type A 200 U injection at Day 1 followed by botulinum toxin Type A 200 U injection > Week 12; injections into detrusor
  Other Names: BOTOX®
  Arms: 1
Biological: botulinum toxin Type A (300U) — botulinum toxin Type A 300 U injection on Day 1 followed by botulinum toxin Type A 300 U injection > Week 12; injections into detrusor
  Other Names: BOTOX®
  Arms: 2
Other: Normal saline (Placebo); botulinum toxin Type A (200U) — Placebo injection on Day 1 followed by botulinum toxin Type A 200 U injection > 12 weeks; injections into detrusor
  Other Names: BOTOX®
  Arms: 3
Other: Normal saline (Placebo); botulinum toxin Type A (300U) — Placebo injection on Day 1 followed by botulinum toxin Type A 300 U injection > Week 12; injections into detrusor
  Other Names: BOTOX®
  Arms: 4

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of botulinum toxin type A in treating overactive bladder in spinal cord injury or multiple sclerosis patients

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence as a result of neurogenic overactive bladder due to spinal cord injury or multiple sclerosis
* Inadequate response to anticholinergic medication used to treat overactive bladder

Exclusion Criteria:

* History or evidence of pelvic or urologic abnormality
* Previous or current diagnosis of bladder or prostate cancer
* Urinary tract infection at time of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (12):
- Middlebury, Connecticut, United States
- Rio de Janeiro, Brazil
- Victoria, British Columbia, Canada
- Salouël, France
- Milan, Italy
- Amsterdam, Netherlands
- Porto, Portugal
- Singapore, Singapore
- Pretoria, South Africa
- Santa Cruz de Tenerife, Spain
- Hualien City, Taiwan
- Scunthorpe, United Kingdom

REFERENCES:
- [Derived] Cuervo J, Castejon N, Khalaf KM, Waweru C, Globe D, Patrick DL. Development of the Incontinence Utility Index: estimating population-based utilities associated with urinary problems from the Incontinence Quality of Life Questionnaire and Neurogenic Module. Health Qual Life Outcomes. 2014 Oct 8;12:147. doi: 10.1186/s12955-014-0147-7. PMID 25288099
- [Derived] Sussman D, Patel V, Del Popolo G, Lam W, Globe D, Pommerville P. Treatment satisfaction and improvement in health-related quality of life with onabotulinumtoxinA in patients with urinary incontinence due to neurogenic detrusor overactivity. Neurourol Urodyn. 2013 Mar;32(3):242-9. doi: 10.1002/nau.22293. Epub 2012 Sep 10. PMID 22965657
- [Derived] Cruz F, Herschorn S, Aliotta P, Brin M, Thompson C, Lam W, Daniell G, Heesakkers J, Haag-Molkenteller C. Efficacy and safety of onabotulinumtoxinA in patients with urinary incontinence due to neurogenic detrusor overactivity: a randomised, double-blind, placebo-controlled trial. Eur Urol. 2011 Oct;60(4):742-50. doi: 10.1016/j.eururo.2011.07.002. Epub 2011 Jul 13. PMID 21798658

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin Type A (300U): botulinum toxin Type A (300U)
- Botulinum Toxin Type A (200U): botulinum toxin Type A (200U)
- Placebo: Normal saline (placebo)
Period: Treatment Cycle 1
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Started | 91 | 92 | 92
Completed | 76 | 80 | 81
Not Completed | 15 | 12 | 11
Period: Treatment Cycle 2
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Started | 63 (32 from the 300U group + 31 from the Placebo group entered Cycle 2) | 74 (42 from the 200U group + 32 from the Placebo group entered Cycle 2) | 0 (Cycle 1 Placebo pts were randomized to receive 300U or 200 U in Cycle 2)
Completed | 58 | 72 | 0
Not Completed | 5 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo | Total
Number analyzed (Participants) | 91 | 92 | 92 | 275
Age, Customized [Number; unit: participants]
  < 40 years | 30 | 31 | 25 | 86
  Between 40 and 64 years | 56 | 55 | 61 | 172
  Between 65 and 74 years | 4 | 5 | 5 | 14
  >= 75 years | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 49 | 155
  Male | 39 | 38 | 43 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Weekly Episodes of Urinary Incontinence
Description: Change from baseline in the weekly frequency of incontinence episodes at Week 6 after the first treatment. Incontinence is defined as involuntary loss of urine as recorded in a patient bladder diary. A negative number change from baseline indicates a reduction in incontinence episodes (improvement).
Time Frame: Baseline, Week 6
Population: Intent-To-Treat, defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Number of Weekly Episodes
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Number analyzed (Participants) | 91 | 92 | 92
Number of Weekly Episodes
  Baseline | 31.2 (18.14) | 32.5 (18.44) | 36.7 (30.67)
  Week 6 | -19.4 (25.67) | -21.8 (18.06) | -13.2 (20.02)

2. Secondary Outcome: Change From Baseline in Maximum Cystometric Capacity (MCC)
Description: Change from baseline in MCC at Week 6. MCC represents the maximum volume of urine the bladder holds. A positive number change from baseline represents an improvement (increase) in maximum volume of urine the bladder holds.
Time Frame: Baseline, Week 6
Population: Intent-To-Treat, defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Milliliters (mL) of urine
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Number analyzed (Participants) | 91 | 92 | 92
Milliliters (mL) of urine
  Baseline | 246.8 (149.06) | 247.3 (147.61) | 249.4 (139.29)
  Week 6 | 157.2 (185.18) | 157.0 (164.75) | 6.5 (144.77)

3. Secondary Outcome: Change From Baseline in Maximum Detrusor Pressure (MDP)
Description: Change from baseline in MDP during the first involuntary detrusor contraction at week 6. MDP represents the maximum pressure (peak amplitude) in the bladder during the first involuntary contraction of the bladder muscle. The greater the negative number change from baseline, the better the improvement.
Time Frame: Baseline, Week 6
Population: Intent-To-Treat, defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Centimeters of water (cm H2O)
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Number analyzed (Participants) | 91 | 92 | 92
Centimeters of water (cm H2O)
  Baseline | 42.1 (33.21) | 51.7 (40.95) | 41.5 (31.17)
  Week 6 | -26.9 (33.17) | -28.5 (47.82) | 6.4 (41.10)

4. Secondary Outcome: Change From Baseline in Total Score on Incontinence Quality of Life (I-QOL) Questionnaire
Description: Change from baseline in I-QOL questionnaire total score at Week 6, as completed by the patient. The I-QOL is a validated, disease-specific quality of life (QOL) questionnaire containing 22 questions designed to measure impact of urinary incontinence on patients' lives. Each question is answered on a 5-point scale (1 = worst QOL, and 5 = best QOL). The scores are totaled over the 22 questions and normalized to a score of 0-100 (0=worst QOL and 100=best QOL). A positive change from baseline represents an improvement.
Time Frame: Baseline, Week 6
Population: Intent-To-Treat, defined as all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Number on a Scale (Score)
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Number analyzed (Participants) | 91 | 92 | 92
Number on a Scale (Score)
  Baseline | 36.32 (18.685) | 37.46 (20.109) | 35.72 (18.656)
  Week 6 | 24.26 (28.981) | 24.43 (25.372) | 11.71 (20.163)

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized AND treated. S(AE)s are displayed for the placebo-controlled treatment Cycle 1.
Arm/Group | Botulinum Toxin Type A (300U) | Botulinum Toxin Type A (200U) | Placebo
Serious Adverse Events (participants affected / at risk) | 18/89 | 17/91 | 23/90
Other Adverse Events (participants affected / at risk) | 70/89 | 63/91 | 52/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (300U) (N=89) | Botulinum Toxin Type A (200U) (N=91) | Placebo (N=90)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 — Event not related to study drug
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Endocarditis enterococcal (Infections and infestations) | 0 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bursa injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urine cytology abnormal (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 2 | 3
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 — Event not related to study drug
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 — Event not related to study drug
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Event not related to study drug
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (300U) (N=89) | Botulinum Toxin Type A (200U) (N=91) | Placebo (N=90)
Constipation (Gastrointestinal disorders) | 6 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 6
Fatigue (General disorders) | 3 | 8 | 1
Pyrexia (General disorders) | 1 | 6 | 3
Urinary tract infection (Infections and infestations) | 57 | 51 | 36
Nasopharyngitis (Infections and infestations) | 6 | 6 | 3
Influenza (Infections and infestations) | 1 | 5 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5
Urinary retention (Renal and urinary disorders) | 28 | 18 | 3
Haematuria (Renal and urinary disorders) | 9 | 5 | 4
Dysuria (Renal and urinary disorders) | 7 | 5 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo